CLINICAL TRIAL: NCT00672841
Title: Randomized Comparison of β-D-Glucan Surveillance With Preemptive Anidulafungin Versus Standard Care for the Management of Invasive Candidiasis in Surgical Intensive Care Unit Patients
Brief Title: β-D-Glucan (BDG) Surveillance With Preemptive Anidulafungin vs. Standard Care for Invasive Candidiasis in Surgical Intensive Care Unit (SICU) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00003161; GA88517X
Record Dates: First submitted 2008-05-04; First posted 2008-05-06 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2012-11

CONDITIONS: Invasive Candidiasis
Keywords: candidemia; invasive candidiasis; preemptive antifungal therapy; surveillance; β-D-Glucan (BDG)
MeSH Terms: conditions — Candidiasis, Invasive; Candidemia | interventions — Anidulafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Standard care/empiric therapy group
  Interventions: Drug: Empiric antifungal therapy based on physician discretion.
- 1 (Experimental): Active surveillance/ preemptive therapy group
  Interventions: Drug: Preemptive Therapy with Anidulafungin

INTERVENTIONS:
Drug: Preemptive Therapy with Anidulafungin — Subjects in the active surveillance arm who develop a single positive β-D-glucan test will receive preemptive anidulafungin intravenously. Preemptive therapy will include a loading dose of 200mg followed by 100mg maintenance therapy once a day. The loading and maintenance doses are derived from the FDA cleared schedule for Invasive Candidiasis and candidemia. Preemptive therapy will continue for 14 days.
  Other Names: Eraxis
  Arms: 1
Drug: Empiric antifungal therapy based on physician discretion. — Patients in the standard care group may receive antifungal prophylaxis and/or treatment at any time based on the discretion of the treating physician.
  Arms: 2

SUMMARY:
This is a single center, prospective, open label assessment of β-D-glucan surveillance with preemptive anidulafungin therapy versus standard care for the prevention of invasive candidiasis in at-risk surgical intensive care unit (SICU) patients. Subjects will be stratified by APACHE II score and randomized in 3:1 fashion to either biweekly surveillance using the β-D-glucan assay or standard care. Subjects in the active monitoring arm will receive intravenous anidulafungin should the β-D-glucan exceed 60 pg/mL on a single determination. Subjects in the standard care arm will have biweekly blood draws for β-D-glucan, but the specimens will be batched and tested retrospectively. Antifungal use in the standard care arm is at the discretion of the treating physicians. The primary study end-points are the feasibility of a preemptive antifungal strategy in a SICU setting, β-D-glucan test characteristics, and the safety and tolerability of preemptive anidulafungin. Risks associated with study participation include the risks associated with blood draws, study drug related side effects, and the potential for loss of confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Admission to the intensive care unit for ≥ 72 hours and expected to stay an additional 48 hours
* IV access for administration of study drug
* Subject (or subject's legal representative) able to give written informed consent

Exclusion Criteria:

* History of hypersensitivity or intolerance to echinocandin antifungals
* Liver function test (ALT, AST (aspartate aminotransferase), and/or total bilirubin) greater than 10 times the upper limits of normal (ULN)
* Pregnant or lactating women
* Treatment with systemic antifungal therapy within the preceding 7 days
* Documented invasive fungal infection at baseline/screening
* Life expectancy less than 2 days or moribund

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-06; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly E Hanson, MD, Principal Investigator — Utah; Barbara D Alexander, MD, Principal Investigator — Duke; John Perfect, MD, Principal Investigator — Duke
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Hanson KE, Pfeiffer CD, Lease ED, Balch AH, Zaas AK, Perfect JR, Alexander BD. beta-D-glucan surveillance with preemptive anidulafungin for invasive candidiasis in intensive care unit patients: a randomized pilot study. PLoS One. 2012;7(8):e42282. doi: 10.1371/journal.pone.0042282. Epub 2012 Aug 6. PMID 22879929

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from June 2008 to December 2010 on three intensive care units.
Groups:
- Standard Care, Empiric Treatment: Standard care group. Empiric antifungal therapy initiated by physician preference for the treatment of suspected invasive candidiasis.
- Active Surveillance, Preemptive Therapy: Active surveillance group. Preemptive therapy (i.e., intravenous anidulafungin 200mg on day one, then 100mg daily x 14 days) initiated in response to a positive 1,3-beta-D glucan test for the presumptive early treatment of invasive candidiasis
Period: Overall Study
Arm/Group | Standard Care, Empiric Treatment | Active Surveillance, Preemptive Therapy
Started | 17 | 47
Completed | 16 | 32
Not Completed | 1 | 15
Not completed — Comfort care | 1 | 4
Not completed — icteric specimens | 0 | 3
Not completed — Antifungal therapy, negative glucan | 0 | 4
Not completed — Adverse Event | 0 | 3
Not completed — Pregnancy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Active Surveillance, Preemptive Therapy: Active surveillance group. Preemptive therapy initiated in response to a positive 1,3-beta-D glucan test for the presumptive early treatment of invasive candidiasis
- Total: Total of all reporting groups
Arm/Group | Standard Care, Empiric Treatment | Active Surveillance, Preemptive Therapy | Total
Number analyzed (Participants) | 17 | 47 | 64
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 30 | 41
  >=65 years | 6 | 17 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (19) | 53 (20) | 53 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 16 | 20
  Male | 13 | 31 | 44
Region of Enrollment [Number; unit: participants]
  United States | 17 | 47 | 64

OUTCOME MEASURES:

1. Primary Outcome: Clinical Utility of Biweekly β-D-glucan (BDG) Testing in At-risk Intensive Care Unit (ICU) Patients.
Description: Clinical utility was defined as β-D-glucan test performance. Biweekly βDG testing used a threshold of ≥ 60 pg/ml to indicate a positive test for invasive candidiasis. True and false positives, and true and false negatives were confirmed using a composite clinical definition of invasive candidiasis that combines physical symptom/signs and microbiology. Cases of proven/probable invasive fungal infection (IFI) were adjudicated by a single reviewer blinded to group assignment and BDG results.
Time Frame: Participants were followed until ICU discharge, an average of 17 days
Population: Two study subjects in the preemptive therapy arm were excluded from the analysis of assay sensitivity and specific due to icteric serum specimens.
Measure: Number; unit: participants
Arm/Group | Active Surveillance, Preemptive Therapy | Standard Care, Empiric Treatment
Number analyzed (Participants) | 45 | 17
participants
  True BDG Positives | 3 | 3
  True BDG Negative | 19 | 9
  False BDG Positives | 23 | 5
  False BGD Negatives | 0 | 0
Statistical Analysis 1: Comparison: Active Surveillance, Preemptive Therapy vs Standard Care, Empiric Treatment; Clinical sensitivity of the BDG test was calculated for both study groups combined; Test type: Superiority or Other; Sensitivity %; Sensitivity = 100 — Sensitivity [1] = (True positives [n=6]/ True positives + False negatives [n=6])
Statistical Analysis 2: Comparison: Active Surveillance, Preemptive Therapy vs Standard Care, Empiric Treatment; Clinical specificity of the BDG test was calculated for the study groups combined; Test type: Superiority or Other; % Specificity; Specificity = 50 — Specificity [0.50]= True negatives [n=28]/ True negatives + False positives [56])

2. Secondary Outcome: Validate Gene Expression Signatures Predictive of IC
Time Frame: Study Completion, an average of 17 days
Population: Data was not collected for this outcome measure.
Arm/Group | Active Surveillance, Preemptive Therapy | Standard Care, Empiric Treatment
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Incidence of Proven or Probable Invasive Fungal Infection (IFI)
Description: Institution specific criteria were used to establish a diagnosis of proven or probable invasive candidiasis. Other IFIs were classified according to the European Organization for Research and Treatment of Cancer/Mycosis Study Group (EORTC/MSG) criteria. However, BDG results were not factored into the EORTC/MSG criteria.
Time Frame: Participants were followed until ICU discharge, an average of 17 days
Population: 4 subjects in the preemptive therapy were excluded from this analysis. These subjects were treated with empiric antifungal therapy despite repeatedly negative glucan results.
Measure: Number; unit: participants
Groups:
- Active Surveillance, Preemptive Therapy: Active surveillance group. Preemptive therapy initiated in response to a positive 1,3-beta-D glucan (BDG) test for the presumptive early treatment of invasive candidiasis
Arm/Group | Standard Care, Empiric Treatment | Active Surveillance, Preemptive Therapy
Number analyzed (Participants) | 17 | 41
participants | 3 | 3
Statistical Analysis 1: Comparison: Standard Care, Empiric Treatment vs Active Surveillance, Preemptive Therapy; The clinic sensitivity of the BDG test was calculated for both study groups combined; Test type: Superiority or Other; Sensitivity; Percent Sensitivity = 100 — Sensitivity = (true positives [n=6]/true positives + false negative [n=6])
Statistical Analysis 2: Comparison: Standard Care, Empiric Treatment vs Active Surveillance, Preemptive Therapy; The clinical specificity of the BDG test was calculated for both study groups combined; Test type: Superiority or Other; Specificity; Percent Specificity = 52 — Specificity [0.52]= (True negatives [n=30]/True negatives + false positives [n=58])

4. Primary Outcome: Safety and Tolerability of Preemptive Anidulafungin
Description: reported as the Number of Adverse Events Possibly Related to Study Drug
Time Frame: weekly until ICU discharge
Population: Subjects receiving at least 1 dose of anidulafungin were assessed.
Measure: Number; unit: events
Arm/Group | Standard Care, Empiric Treatment | Active Surveillance, Preemptive Therapy
Number analyzed (Participants) | 17 | 45
events | 0 | 10

ADVERSE EVENTS:
Arm/Group | Standard Care, Empiric Treatment | Active Surveillance, Preemptive Therapy
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/47
Other Adverse Events (participants affected / at risk) | 0/17 | 10/47
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Standard Care, Empiric Treatment (N=17) | Active Surveillance, Preemptive Therapy (N=47)
Thrombocytopenia (Blood and lymphatic system disorders) | 0/5 (0) | 2/21 (2)
Abnormal liver function tests (Hepatobiliary disorders) | 0/5 (0) | 9/21 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 0/5 (0) | 2/21 (2)

LIMITATIONS AND CAVEATS:
This study represents a 1st attempt at preemptive antifungal therapy based on the fungal biomarker 1,3-Beta-D-Glucan in the intensive care unit. Main limitation: the small number of subjects with proven/probable invasive candidiasis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No